CLINICAL TRIAL: NCT01179178
Title: A Dangerous Triad in Ageing and in COPD - Reduced Muscle Mass, Impaired Muscle Function and Malnutrition
Brief Title: A Dangerous Triad in Ageing and in Chronic Obstructive Pulmonary Disease (COPD) - Reduced Muscle Mass, Impaired Muscle Function and Malnutrition
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government); The Swedish Heart and Lung Association (Other); Swedish Heart Lung Foundation (Other)
Other Study IDs: UGOTTriad; Grant (Other Grant/Funding Number: The Swedish Research Council 2006-3320)
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2006-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD-patients
- Older adults (65-81 y)

SUMMARY:
The investigators have taken part in the development of simple muscle function tests and studied physical training and energy turnover in patients with chronic obstructive pulmonary disease, COPD. The investigators have found that muscle wasting in COPD is related to poor prognosis and that physical training might lead to improved, less energy-demanding muscle function. Elderly subjects also suffer from muscle wasting that leads to frailty, poor autonomy and, secondarily, fractures. In the planned study the investigators will validate simple muscle function tests (hand grip strength, heel rise test, voluntary quadriceps muscle strength, 30 m walking test and balance tests) in both groups by relating them to an involuntary, magnet stimulated, test of quadriceps force, HRQL, tests of body composition (impedance, DXA) and recordings of physical activity. The relation between food intake, systemic inflammation, muscle mass and function will be analysed.

The study has been ethically approved and started in COPD patients and will be expanded to a representative sample of elderly.

Simple, evaluated muscle function tests applied in primary care may be used for early detection of muscle dysfunction in COPD patients and elderly so that early intervention against impaired muscle function can be started. Analyses of food intake and of inflammatory markers might identify factors of special importance for muscle dysfunction, which eventually might lead to improved dietary therapy and pharmacological interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between 65 and 81 years of age, randomly selected from the national registration, are invited to take part in the study.
* Patients referred to the outpatient clinic of the lung unit at Sahlgrenska University Hospital with a diagnosis of COPD are asked for participation.
* Inclusion criteria for COPD patients:
* Clinical diagnosis of COPD
* FEV% < normal value minus 2 SD
* Smoking history; 10 pack years or more

Exclusion Criteria:

* Any specific muscular disease
* Severe disease or handicap making investigations impossible
* Exclusion criteria for COPD patients:
* Any specific muscular disease
* Any co-existing serious disease

Ages: 65 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Outpatients (COPD) and older adults living in Gothenburg
Sampling Method: Probability Sample
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Clinical Nutrition, Sahlgrenska Academy at University of Gothenburg, Gothenburg, Sweden